CLINICAL TRIAL: NCT01111526
Title: A Phase I/II Trial Evaluating the Use of Histone Deacetylase Inhibitor LBH589 in Addition to Corticosteroids in Patients With Acute Graft Versus Host Disease
Brief Title: Histone Deacetylase Inhibitor LBH589 in Addition to Corticosteroids in Patients With Acute Graft Versus Host Disease (GVHD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15618; CLBH589BUS20T (Other: Novartis)
Record Dates: First submitted 2010-04-16; First posted 2010-04-27 (Estimated); Results first posted 2016-12-22 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2016-08

CONDITIONS: Graft-Versus-Host Disease
Keywords: Graft versus host disease; GVHD; allogeneic transplant; acute GVHD; chronic GVHD
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LBH589, in Addition to Glucocorticoids (Experimental): Phase I Dose Escalation, Followed by Phase II Treatment at Maximum Tolerated Dose (MTD) of LBH589, in Addition to Glucocorticoids.
  Interventions: Drug: Panobinostat (LBH589)

INTERVENTIONS:
Drug: Panobinostat (LBH589) — Phase I Initial Treatment Plan - Intravenous (IV) Formulation: Up to 4 dose levels (DL) of LBH589 IV formulation to establish LBH589 Maximum Tolerated Dose (MTD) in acute GVHD treatment. The first 4 participants began this treatment plan, before the IV Formulation became unavailable.
  DL -1: 1.25 mg/m^2 IV; DL 1: 2.5 mg/m^2 IV; DL 2: 5 mg/m^2 IV; DL 3: 7.5 mg/m^2 IV; DL 4: 10 mg/m^2 IV.
  Phase I Revised Treatment Plan - Oral Formulation (to replace IV Formulation): Dose escalation levels for LBH589; participants treated with LBH589 by mouth (PO) 3 times a week (48 hours apart) every week for 4 weeks.
  DL -1: 5 mg PO; DL 1: 10 mg PO (starting dose level); DL 2: 15 mg PO; DL 3: 20 mg PO; DL 4: 25 mg PO.
  Phase II Treatment Plan: LBH589 PO at MTD, 3 times a week (48 hours apart) every week for 4 weeks.

SUMMARY:
To test a new agent, LBH589, in combination with glucocorticoids as initial therapy of acute graft versus host disease (GVHD).

DETAILED DESCRIPTION:
Dose escalation study to test the safety (Phase I), pharmacology and preliminary clinical activity (Phase II) of a Novel histone deacetylase (HDAC) inhibitor, LBH589, in the treatment of the following GVHD presentations: Classic, Late-onset acute GVHD, Recurrent acute GVHD, Overlap syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients receiving allogeneic hematopoietic cell transplantation (HCT) with peripheral blood, bone marrow or cord blood stem cells regardless of initial diagnosis who develop a clinical diagnosis of acute GVHD as defined in Section 2 diagnosed and treated with systemic glucocorticoids within 72 hours prior to enrollment. Biopsy of involved skin and gastrointestinal tract is strongly encouraged, but not required for study entry. For patients with aspartic transaminase (AST) or alanine transaminase (ALT) or Alkaline phosphatase with gamma-glutamyltransferase (GGT) elevations without bilirubin elevation must have a liver biopsy to document GVHD diagnosis. Patients should meet one of the following criteria:

   If GVHD is present in an isolated organ:
   1. Skin rash involvement of a minimum of 50% of body surface area in absence of documented drug allergy or infectious etiology.
   2. Diarrhea with a minimum stool volume of 500 mL/day and/or a minimum of 2 stools above baseline/day in absence of enterocolitis from C. difficile or other documented pathogens.
   3. Increase in bilirubin above upper limit of normal (ULN) in absence of clinically defined veno-occlusive disease.
   4. Isolated increased AST and/or ALT and/or increased alkaline phosphatase above ULN with GGT elevation above ULN with documented liver GVHD biopsy.

   If GVHD presentation involves >/= 2 organs: GVHD Grade >/= II as defined in Table D of protocol.
2. Male or female patients aged 18 or older at time of enrollment
3. Signed informed consent
4. Absolute neutrophil count (ANC) greater than 500/μL, platelets >/= 20 x 10^9/L supported by platelet transfusion and hemoglobin >/= 8 g/dl supported by red cell transfusion.
5. Calculated creatinine clearance (CrCl) >/= 30 mL/min (MDRD Formula)
6. Serum potassium >/= lower limit of normal (LLN), Total serum calcium [corrected for serum albumin] or ionized calcium >/= LLN, Serum magnesium >/= LLN and Serum phosphorus >/= LLN on the day of LBH589 administration
7. Thyroid-stimulating hormone (TSH) </= ULN and free T4 within normal limits at the time of patient enrollment within baseline laboratories. Patients are permitted to receive thyroid hormone replacement to treat underlying hypothyroidism
8. Baseline multiple gated acquisition scan (MUGA) or echocardiogram (ECHO) must demonstrate left ventricular ejection fraction (LVEF) >/= the lower limit of the institutional normal before transplantation.

Exclusion Criteria:

1. Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not using an effective method of birth control. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months). Women of childbearing potential must have a negative serum pregnancy test within 24 hrs of receiving the first dose of study medication if a pregnancy test was not done pre-transplant. Male patients whose sexual partners are WOCBP not using effective birth control
2. Patients requiring mechanical ventilation support.
3. Active, uncontrolled life threatening viral or fungal disease, such as cytomegalovirus (CMV) pneumonia or gastroenteritis, Aspergillus pneumonia or brain abscess. For bacterial or viral infections, patients must be receiving therapy and have no signs of progression for 48 hours prior to enrollment. For fungal infection patients must be receiving systemic anti-fungal therapy and have no signs of progression for 1 week prior to enrollment. Progressing infection is defined as hemo-dynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infections. Persisting fever without other signs of symptoms will not be interpreted as progressing infections.
4. Receipt of other investigational new drugs for GVHD including agents used for GVHD prophylaxis within 30 days. The following agents are not considered experimental and therefore are not excluded: cyclosporine, tacrolimus, sirolimus, glucocorticoids, antithymocyte globulin, replacement corticosteroid therapy for hypoadrenalism and methotrexate.
5. HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer within 30 days.
6. Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first LBH589 treatment.
7. Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

   1. Patients with congenital long QT syndrome.
   2. History or presence of sustained ventricular tachyarrhythmia. (Patients with a history of a controlled atrial arrhythmia are eligible).
   3. Any history of ventricular fibrillation or torsade de pointes.
   4. Bradycardia defined as heart rate (HR)< 50 bpm. Patients with pacemakers are eligible if HR >/= 50 bpm.
   5. Patients are excluded if the average of the QT Corrected by the Fridericia Formula (QTcF) is > 470 msec on the screening EKGs.
   6. Right bundle branch block + left anterior hemiblock (bifascicular block).
   7. Patients with myocardial infarction or unstable angina </= 6 months prior to starting study drug.
   8. Other clinically significant heart disease (e.g., congestive heart failure (CHF) New York Heart Association class III or IV, or uncontrolled hypertension.
8. Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug.
9. Concomitant use of CYP3A4 inhibitors with the exception of tacrolimus, voriconazole (or posaconazole), cyclosporine that are required for all GVHD patients to control GVHD and prevent mould infections (Appendix A of protocol).
10. Patients with known positivity for human immunodeficiency virus (HIV) before transplant.
11. Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-04; Primary Completion 2015-10 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lia Perez, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: H. Lee Moffitt Cancer Center & Research Institute — http://www.moffitt.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center, September 2010 through December 2014.
Groups:
- Phase I Participants Not Evaluable for MTD: Participants who began treatment before the formulation change.
- Phase I Participants Evaluable for MTD: Participants treated after the formulation change.
- Phase II Participants Treated at MTD: All participants enrolled during Phase II.
Period: Overall Study
Arm/Group | Phase I Participants Not Evaluable for MTD | Phase I Participants Evaluable for MTD | Phase II Participants Treated at MTD
Started | 4 | 8 | 10
Completed | 4 | 7 | 8
Not Completed | 0 | 1 | 2
Not completed — GVHD Disease Progression | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: All participants. All participants received study treatment.
Arm/Group | LBH589, in Addition to Glucocorticoids
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 55 [34 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) in Milligrams
Description: MTD of LBH589 in addition to glucocorticoids as treatment for Graft Versus Host Disease (GVHD) manifestations. MTD in Milligrams (mg), taken by mouth (PO), 3 times per week, for 4 weeks. The oral formulation replaced the IV formulation (which became unavailable) after the first 4 participants were treated. Dose limiting toxicity (DLT) is defined by the occurrence of Common Toxicity Criteria (CTC) grade 3 or greater toxicity that is unexpected with transplantation, except for hematological toxicity, where DLT is defined as absolute neutrophil count (ANC) <750, and for those participants who were platelet transfusion independent is defined as platelets <10 K.
Time Frame: 2 years, 8 months
Population: All participants treated with Oral Formulation LBH589, during Phase I Dose Escalation.
Measure: Number; unit: MTD of oral LBH589 in milligrams
Arm/Group | LBH589, in Addition to Glucocorticoids
Number analyzed (Participants) | 8
MTD of oral LBH589 in milligrams | 5

2. Primary Outcome: Phase II: Overall Rate of Response (ORR)
Description: Rate of Complete Response (CR), Partial Response (PR), Progressive Disease (PD) and Stable Disease (SD). Assessment of GVHD will include the skin, liver and gut. Other possible etiologies of organ disease such as C difficile enterocolitis, viral infection, drug reaction, veno-occlusive disease of the liver, etc., will be excluded by appropriate tests. CR is defined as resolution of GVHD in all evaluable organs with no subsequent additional treatment given for acute GVHD. PR is defined as improvement in ≥ one evaluable organ without deterioration in at least one other. PD is defined as deterioration in at least on evaluable organ. SD is defined as the absence of any difference sufficient to meet minimal criteria for improvement or deterioration in any evaluable organs.
Time Frame: 1 year, 2 months
Population: All participants treated at maximum tolerated dose (MTD) of Oral Formulation LBH589, and evaluable at planned time of analysis.
Measure: Number; unit: participants
Arm/Group | LBH589, in Addition to Glucocorticoids
Number analyzed (Participants) | 16
participants
  Complete Response | 13
  Partial Response | 2
  Progressive Disease | 1
  Stable Disease | 0

3. Secondary Outcome: Incidence of GVHD Flares Requiring Increasing Immune Suppressive Therapy
Description: Number of participants with GVHD flares requiring increasing immune suppressive therapy within 36 days of study initiation. Cumulative incidence of GVHD flares requiring increasing immune suppressive therapy will be analyzed using the competing risk method by Gray (1988). GVHD flares (progressive disease (PD)) may result in discontinuation from Panobinostat.
Time Frame: Up to 36 days per participant
Population: All participants that received Oral Formulation LBH589 at MTD (5 mg) 3 times per week, for 4 weeks.
Measure: Number; unit: participants
Arm/Group | LBH589, in Addition to Glucocorticoids
Number analyzed (Participants) | 16
participants | 1

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) at one year post initiation of therapy.
Time Frame: 1 year
Population: All participants that received Oral Formulation LBH589 at MTD (5 mg) 3 times per week, for 4 weeks.
Measure: Number; unit: participants
Arm/Group | LBH589, in Addition to Glucocorticoids
Number analyzed (Participants) | 16
participants
  OS at 1 year | 11
  Death before 1 year: sepsis | 1
  Death before 1 year: relapse | 2
  Death before 1 year: GVHD | 1
  Death before 1 year: Cardiogenic shock | 1

5. Secondary Outcome: Occurrence of Discontinuation of All Immune Suppression
Description: Number of participants discontinuing all immune suppression without subsequent flare by 1 year post initiation of therapy.
Time Frame: 1 year
Population: All participants that received Oral Formulation LBH589 at MTD (5 mg) 3 times per week, for 4 weeks and were evaluable at 365 days.
Measure: Number; unit: participants
Arm/Group | LBH589, in Addition to Glucocorticoids
Number analyzed (Participants) | 11
participants | 0

6. Secondary Outcome: Chronic GVHD Onset
Description: Chronic GVHD onset in participants without overlap syndrome at initiation of study therapy. Number of participants with overlap syndrome at MTD.
Time Frame: Up to 1 year
Population: All participants that received Oral Formulation LBH589 at MTD (5 mg) 3 times per week, for 4 weeks.
Measure: Number; unit: participants
Arm/Group | LBH589, in Addition to Glucocorticoids
Number analyzed (Participants) | 16
participants | 6

7. Secondary Outcome: Chronic GVHD Severity at MTD
Description: Chronic GVHD maximum severity grade at MTD, in participants without overlap syndrome at initiation of study therapy. Maximum c-GVHD severity: Mild, Moderate, Severe.
Time Frame: Up to 1 year
Population: All participants that received Oral Formulation LBH589 at MTD (5 mg) 3 times per week, for 4 weeks, had overlap syndrome at MTD and were evaluable at time of analysis.
Measure: Number; unit: participants
Arm/Group | LBH589, in Addition to Glucocorticoids
Number analyzed (Participants) | 5
participants
  Mild | 2
  Moderate | 1
  Severe | 1

8. Secondary Outcome: Stable or Improved Chronic GVHD Severity Score
Description: Stable or improved Chronic GVHD score: Improved Mild to None; Improved Severe to Moderate; Improved Moderate to None, Remained Stable at Mild.
Time Frame: 1 year
Population: All participants that received Oral Formulation LBH589 at MTD (5 mg) 3 times per week, for 4 weeks, had overlap syndrome at MTD and were evaluable at 1 year.
Measure: Number; unit: participants
Arm/Group | LBH589, in Addition to Glucocorticoids
Number analyzed (Participants) | 5
participants
  Improved: Mild to None | 1
  Improved: Severe to Moderate | 1
  Improved: Moderate to None | 1
  Stable: Remained Stable at Mild | 1

9. Secondary Outcome: Occurrence of Possibly Related Adverse Events
Description: Number of participants with adverse events possibly related to study treatment, per event category.
Time Frame: 5 years, 3 months
Population: All participants
Measure: Number; unit: participants
Arm/Group | LBH589, in Addition to Glucocorticoids
Number analyzed (Participants) | 22
participants
  Thrombocytopenia | 11
  Leukopenia | 6
  Anemia | 2
  Hypertriglyceridemia | 5
  Hypercholesterolemia | 3
  Fatigue | 1
  Hepatobiliary disorders | 1

ADVERSE EVENTS:
Time Frame: 5 years, 3 months
Description: All participants. All events are listed regardless of causality.
Arm/Group | LBH589, in Addition to Glucocorticoids
Serious Adverse Events (participants affected / at risk) | 11/22
Other Adverse Events (participants affected / at risk) | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LBH589, in Addition to Glucocorticoids (N=22)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac disorders - Other, Hypotension (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Gastrointestinal disorders - Other, severe diarrhea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, GVHD/VOD (Gastrointestinal disorders) | 1 (2)
Gastrointestinal disorders - Other, Severe GVHD (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disorders - Other, suspected drug toxicity to liver (Hepatobiliary disorders) | 1 (1)
Infections and infestations - Other, cellulitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Renal and urinary disorders - Other, put on dialysis (Renal and urinary disorders) | 1 (1)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LBH589, in Addition to Glucocorticoids (N=22)
Platelet count decreased (Investigations) | 19 (43)
White blood cell decreased (Investigations) | 12 (21)
Cholesterol high (Investigations) | 11 (17)
Alkaline phosphatase increased (Investigations) | 5 (5)
Neutrophil count decreased (Investigations) | 5 (6)
Blood bilirubin increased (Investigations) | 3 (3)
Alkaline aminotransferase increased (Investigations) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Hypertension (Vascular disorders) | 16 (35)
Hypotension (Vascular disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 14 (36)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 7 (10)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Cardiac disorders - Other, cardiac arrhythmia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (4)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cardiovascular toxicity (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The discontinuation of the IV Formulation of LBH589 required a treatment plan change to Oral Formulation LBH589, after the first 4 participants were treated. The study accrued fewer participants than investigators had planned to evaluate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes